CLINICAL TRIAL: NCT00755638
Title: A Randomized, Double-Blind, Placebo-Controlled, Single-Dose, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Effects of ACE-031 (ActRIIB-IgG1) in Healthy, Postmenopausal Volunteers
Brief Title: A Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study of ACE-031 (ActRIIB-IgG1)in Healthy Postmenopausal Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Niels Borgstein, MD, Acceleron Pharma Inc.
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: A031-01
Record Dates: First submitted 2008-09-17; First posted 2008-09-19 (Estimated); Last update posted 2009-07-14 (Estimated); Status verified 2009-07

CONDITIONS: Muscle Loss
MeSH Terms: conditions — Muscular Atrophy | interventions — ACVR2B protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- single (Experimental): 8 subjects (6 active and 2 placebo)
  Interventions: Biological: ACE-031

INTERVENTIONS:
Biological: ACE-031 — single subcutaneous dose of ACE-031

SUMMARY:
Single center, randomized, single dose study to evaluate the safety, tolerability, pharmacokinetic and pharmacodynamic effects of ACE-031 in healthy postmenopausal volunteers

ELIGIBILITY:
Key Inclusion Criteria:

1. Subject is a postmenopausal woman, 45-75 years old (inclusive)
2. Subject has a body mass index (BMI) of > 18.5 to < 30
3. Subject must give written informed consent

Key Exclusion Criteria:

1. Subject has a history of malignancy. However, a subject with a history of excised or treated basal cell carcinoma, cervical carcinoma in-situ, or less than or equal to 2 squamous cell carcinomas is eligible to participate in this study.
2. Subject has a history of clinically significant (as determined by the Investigator) cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease.
3. Subjects with chronic stable diseases including migraines, hypertension, hyperthyroid disorder, hypothyroid disorder, gastroesophageal reflux disease, or mild depression/anxiety will be excluded unless the investigator does not have safety or compliance concerns at study entry.
4. Subject has a history of opportunistic infection (e.g. invasive candidiasis or pneumocystis pneumonia).
5. Subject has had a serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., septicemia) within the 3 months prior to screening.
6. Subject has a history of severe allergic or anaphylactic reactions.
7. Subject had surgery within the previous 3 months (other than minor cosmetic surgery or minor dental procedures).
8. Subject had a fever (body temperature > 38°C) or symptomatic viral or bacterial infection within 2 weeks prior to dosing.
9. Subject has a positive Tuberculin skin test (Mantoux)
10. Subject has a history of hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV), or human immunodeficiency virus (HIV).
11. Subject has a recent or clinically significant history of drug or alcohol abuse, or tests positive in a urine screen for alcohol or drugs of abuse.
12. Subject consumed any alcohol within 48 hours prior to dosing.
13. Subject has donated or lost ≥ 499 mL of whole blood within 56 days prior to study drug administration.
14. Subject has taken any hormone replacement therapy within 3 months prior to study enrollment, or plans to begin hormone replacement therapy at any time during the study.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of single, escalating doses of ACE-031 in healthy postmenopausal volunteers | specified timepoints in the protocol

SECONDARY OUTCOMES:
To estimate the pharmacokinetic (PK) and pharmacodynamic (PD) effects of ACE-031 | specified timepoints in the protocol

CONTACTS AND LOCATIONS:
Locations (1):
- Acceleron Investigative Site, Montreal, Quebec, Canada